CLINICAL TRIAL: NCT00433862
Title: Molecular Changes and Biomarkers in Chronic Myeloproliferative Disorders
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070090; 07-CC-0090
Record Dates: First submitted 2007-02-09; First posted 2007-02-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-19

CONDITIONS: Polycythemia Vera; Essential Thrombocytosis; Idiopathic Myelofibrosis; Neutrophils; Chronic Myeloproliferative Disorders
Keywords: Polycythemia Vera; Essential Thrombocytosis; Idiopathic Myelofibrosis; Janus Kinase 2; CD177; Chronic Myeloproliferative Disorders; PV; Essential Thrombocythemia; ET; IM
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis; Myeloproliferative Disorders

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The three main chronic myeloproliferative disorders are polycythemia vera (PV), essential thrombocythemia (ET) and idiopathic myelofibrosis (IMF). These are clonal neoplastic diseases characterized by proliferation of one or more hematopoietic lineages. Recently a mutation of the Janus Kinase 2 (JAK2) gene that leads to the substitution of phenylalanine for valine at position 617 of the JAK2 protein, JAK2 V617F, has been found in 76% to 97% of patients with PV, 29% to 57% of patients with ET and 50% of patients with IMF. This mutation confers constitutive activity on to the JAK2 protein and appears to play an important role in the pathobiology of these conditions. However, not all patients with myeloproliferative disorders have this mutation and it may not be the primary cause of these diseases. The primary goal of this prospective natural history study is to investigate the molecular basis of these diseases in groups of patients who have JAK2 V617F and in those who do not. A second goal is to identify biomarkers for PV and the other myeloproliferative disorders that are easier to measure than JAK2 V617F. Approximately, 150 patients with myeloproliferative disorders will be studied over 3 years. The studies will involve the collection of 40 mL to 50 mL of peripheral blood from each subject. The blood will be used to assess neutrophil gene and protein expression, gene polymorphisms, and plasma protein levels.

DETAILED DESCRIPTION:
The three main chronic myeloproliferative disorders are polycythemia vera (PV), essential thrombocythemia (ET) and idiopathic myelofibrosis (IMF). These are clonal neoplastic diseases characterized by proliferation of one or more hematopoietic lineages. Recently a mutation of the Janus Kinase 2 (JAK2) gene that leads to the substitution of phenylalanine for valine at position 617 of the JAK2 protein, JAK2 V617F, has been found in 76% to 97% of patients with PV, 29% to 57% of patients with ET and 50% of patients with IMF. This mutation confers constitutive activity on to the JAK2 protein and appears to play an important role in the pathobiology of these conditions. However, not all patients with myeloproliferative disorders have this mutation and it may not be the primary cause of these diseases. The primary goal of this prospective natural history study is to investigate the molecular basis of these diseases in groups of patients who have JAK2 V617F and in those who do not. A second goal is to identify biomarkers for PV and the other myeloproliferative disorders that are easier to measure than JAK2 V617F. Approximately, 150 patients with myeloproliferative disorders will be studied over 3 years. The studies will involve the collection of 40 mL to 50 mL of peripheral blood from each subject. The blood will be used to assess neutrophil gene and protein expression, gene polymorphisms, and plasma protein levels.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Diagnosis or suspected diagnosis of PV, ET, or IMF. The World Health Organization Criteria will be used for diagnosing this disorder. In brief, the criteria for PV is hemoglobin greater than 18.5 g/dL in men and greater than 16.5 g/dL in women and splenomegaly on palpation in the absence of secondary erythrocytosis. If splenomegaly is absent, the patient must have 2 of the following 4 minor criteria: platelet count greater than 400 x 10(9)/L, leukocyte count greater than 12 x 10(9)/L, marrow biopsy with trilineage increase in cellularity, and low serum erythropoietin level. The criteria for EF is a platelet count greater than 600 x 10(9)/L with no known cause of reactive thrombocytosis and a normal hemoglobin. The criteria for IMF is fibrosis of the bone marrow and splenomegaly without preceding PV, ET or chronic myelogenous leukemia.
  2. Both male and female subjects will be studied.
  3. Any ethnic group.
  4. 18 years of age or older.

EXCLUSION CRITERIA:

Subjects will be excluded if they have any of the following conditions:

1. Increased blood counts due to a disease other than chronic myeloproliferation.
2. Know history of anemia (hematocrit less than 12.0 mg/dL).
3. Pregnancy.
4. Infection with HIV, hepatitis B, or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-02-06; Study Completion 2010-05-19

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - VA Medical Center, Washington D.C., Washington D.C., District of Columbia
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] DAMESHEK W. Some speculations on the myeloproliferative syndromes. Blood. 1951 Apr;6(4):372-5. No abstract available. PMID 14820991
- [Background] Spivak JL. Polycythemia vera: myths, mechanisms, and management. Blood. 2002 Dec 15;100(13):4272-90. doi: 10.1182/blood-2001-12-0349. Epub 2002 Aug 8. No abstract available. PMID 12393615
- [Background] el-Kassar N, Hetet G, Briere J, Grandchamp B. Clonality analysis of hematopoiesis in essential thrombocythemia: advantages of studying T lymphocytes and platelets. Blood. 1997 Jan 1;89(1):128-34. PMID 8978285